CLINICAL TRIAL: NCT04013035
Title: The Impact of Fetal Viability and Cervical Length on Pregnancy Termination Outcomes in Nulliparous Second Trimester Pregnancies
Brief Title: Cervical Length on Pregnancy Termination
Status: Completed | Type: Observational
Sponsor: Kanuni Sultan Suleyman Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Pınar Kadirogulları, principal investigator, M.D, Department of Obstetrics and Gynecology, Kanuni Sultan Suleyman Training and Research Hospital
Other Study IDs: 2015.01.01
Record Dates: First submitted 2019-07-07; First posted 2019-07-09 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Pregnancy Loss
Keywords: Cervix; Length; Viability; prostaglandin; Termination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: cervical length measurement — cervical length measurement at second trimester pregnancy termination in nulliparous pregnant women.

SUMMARY:
Cervical length is used as a parameter to predict cervical insufficiency and onset of labor. However, its role in predicting abortion induction is unclear.To investigate the impact of cervical length measurement and fetal viability on second trimester pregnancy termination duration in nulliparous pregnant women.

DETAILED DESCRIPTION:
Cervical length and fetal viability were evaluated prior to second trimester pregnancy termination due to various indications. nulliparous pregnant women through 13 and 26 gestational weeks in whom pregnancy termination was conducted within 72 hours after admission were included in the study. The subjects were grouped into two groups according to fetal viability.

ELIGIBILITY:
Inclusion Criteria:

-Nulliparous pregnant women at 13-26 weeks of gestation

Exclusion Criteria:

* Patients with multiple gestations,
* multiparous patients or
* patients that had uterine gynecologic surgery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Nulliparous pregnant women at 13-26 weeks of gestation will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
cervical length measurement | 2 days
  cervical length measurement at second trimester pregnancy termination in nulliparous pregnant women. The measurements will be saved as a number in cm.

CONTACTS AND LOCATIONS:
Locations (1):
- Kanuni Sultan Süleyman Training and Research Hospital, Istanbul, Turkey (Türkiye)